CLINICAL TRIAL: NCT00510393
Title: The DESTINY Trial: a Prospective Randomized Multicenter Trial Comparing the Implant of a Drug Eluting Stent (XIENCE V, Abbott Vascular) vs. a Bare Metal Stent (MULTILINK VISION, Abbott Vascular) in the Critically Ischemic Lower Leg
Brief Title: Drug Eluting Stents In The Critically Ischemic Lower Leg
Acronym: DESTINY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Flanders Medical Research Program (FMRP), Flanders Medical Research Program (FMRP)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMRP-002
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: Critical Limb Ischemia; CLI; Drug Eluting Stent; DES; Bare Metal Stent; BMS
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): drug eluting stent
  Interventions: Device: XIENCE V everolimus eluting coronary stent system
- 2 (Placebo Comparator): Bare Metal Stent
  Interventions: Device: MULTILINK VISION coronary stent system

INTERVENTIONS:
Device: XIENCE V everolimus eluting coronary stent system
  Arms: 1
Device: MULTILINK VISION coronary stent system
  Arms: 2

SUMMARY:
The Destiny trial compares the use of bare metal stent systems with drug eluting stent systems in the treatment of infrapopliteal lesions in patients with Critical Limb Ischemia. It will be investigated whether there is a difference in 12 month angiographic patency of the stented area using the 2 different stent systems.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic (> 50%) or occlusive atherosclerotic disease of the infrapopliteal arteries
* A maximum of two focal target lesions in one or more infrapopliteal vessels
* Length of lesion is maximally 40 mm, allowing maximally 2 stents to be implanted
* Reference vessel diameter should be 2-3.5 mm
* Symptomatic critical limb ischemia (Rutherford 4, 5)
* The patient must be > 18 years of age
* Life-expectancy of more than 12 months
* The patient has no child bearing potential or negative serum pregnancy test within 7 days of the index procedure
* The patient must be willing and able to return to the appropriate follow-up times for the duration of the study
* The patient must provide written patient informed consent that is approved by the ethics committee

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for available stent design.
* Unsuccessfully treated (>30% residual stenosis) proximal inflow limiting arterial stenosis
* Untreatable lesion located at the distal outflow arteries
* More than two infrapopliteal lesions in the same limb
* Previously implanted stent(s) or PTA at the same lesion site
* Lesion location requiring kissing stent procedure
* Lesion lies within or adjacent to an aneurysm
* Inflow-limiting arterial lesions left untreated
* The patient has a known allergy to heparin, Aspirin or other anticoagulant/anti-platelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient takes Phenprocoumon (Marcumar).
* The patient has a history of prior life-threatening contrast media reaction.
* The patient is currently enrolled in another investigational device or drug trial.
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* The patient is mentally ill or retarded.
* Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Subject is receiving or scheduled to receive anticancer therapy for malignancy within 30 days prior to or after the procedure
* Subject is receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.) The patient should also not receive inhibitors of CYP3A (such as Itraconazole, and Erythromycin), or inducers of CYP3A (such as Rifampin) within 90 days following the procedure.
* Subject is receiving or is scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Angiographic patency, defined as angiographic binary in-stent restenosis rate (>50% stenosis). | one year

SECONDARY OUTCOMES:
Technical success defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex ultrasound (US) imaging. | procedure
Primary patency rate at each follow-up. Patients that did not receive any BTK-reintervention and do not exhibit significant restenosis on duplex (PVR ≥ 2.4) are defined as being primary patent at the given follow-up. | one year
Limb-salvage rate (LSR) defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot). | one year
Clinical events defined as fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization. | one year
Clinical success defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius, Dendermonde, Belgium; Dierk Scheinert, MD, Principal Investigator — Herzzentrum, Leipzig, Germany
Locations (5):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
- Polyclinique Les Fleurs, Ollioules, France
- Germany (2):
  - Herz-zentrum Bad Krozingen, Bad Krozingen
  - Herzzentrum, Leipzig

REFERENCES:
- [Derived] Bosiers M, Scheinert D, Peeters P, Torsello G, Zeller T, Deloose K, Schmidt A, Tessarek J, Vinck E, Schwartz LB. Randomized comparison of everolimus-eluting versus bare-metal stents in patients with critical limb ischemia and infrapopliteal arterial occlusive disease. J Vasc Surg. 2012 Feb;55(2):390-8. doi: 10.1016/j.jvs.2011.07.099. Epub 2011 Dec 14. PMID 22169682